CLINICAL TRIAL: NCT06755229
Title: Does Smoking Affect the Onset and Duration of Ultrasound-guided Infraclavicular Brachial Plexus Block?
Brief Title: Impact of Smoking on Ultrasound-Guided Infraclavicular Brachial Plexus Block Onset and Duration
Status: Not yet recruiting | Type: Observational
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Mehmet SARGIN, Associate Professor, Selcuk University
Other Study IDs: 2024-12-2
Record Dates: First submitted 2024-12-19; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Smoking, Cigarette; Regional Anesthesia
MeSH Terms: conditions — Cigarette Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-smoker: Never smoked in their life
- Smoker: ≥20 cigarettes/day for>1 year

SUMMARY:
The present study will be conducted involving 40 patients aged 18-65 years with ASA physical status I and II, scheduled for acute or elective hand or forearm surgery under the lateral infraclavicular block. Patients will be divided into two groups based on smoking status: Group I (non-smokers) and Group II (smokers who smoke ≥20 cigarettes/day for over 1 year).

Using a high-frequency linear ultrasound transducer, the axillary artery, vein, and the three nerve cords will be identified in the lateral infraclavicular region. After disinfection with ethanol-chlorhexidine, a sterile drape will be placed, and the attending anesthesiologist will perform the ultrasound-guided infraclavicular brachial plexus block with a triple injection technique. A total of 10 mL of bupivacaine 0.25% and prilocaine 0.05% will be injected at all three nerve cords.

The primary outcome will be the sensory blockade onset time, while secondary outcomes will include the duration of sensory and motor blockade, motor blockade onset time, time to first postoperative rescue analgesia, and total consumption of rescue analgesia. Postoperative pain will be assessed using the Visual Analogue Scale (VAS) within the first 24 hours at intervals of 2, 4, 8, 12, 16, and 24 hours. If VAS exceeds 30 cm, rescue analgesia with 0.05 mg/kg intravenous morphine sulfate will be administered.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I and II
* Scheduled for acute or elective hand or forearm surgery under the lateral infraclavicular block

Exclusion Criteria:

* morbid obesity (body mass index > 40)
* bleeding disorder
* coagulopathy
* medication with vitamin K antagonists
* high-dose or fractionated heparin treatment
* allergy to local anaesthetics
* infection at the site of needle insertion
* peripheral neurological disease
* pregnancy

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 to 65 years, classified as ASA physical status I and II, scheduled for acute or elective hand or forearm surgery with a lateral infraclavicular block.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-03-20 (Estimated)

PRIMARY OUTCOMES:
Sensory blockade onset time | During procedure
  The sensory blockade onset time will be evaluated using a cold ice pack.

SECONDARY OUTCOMES:
Duration of sensory blockade | up to 24 hours
  The duration of sensory blockade will be evaluated as the time between the onset of the sensory block and the complete disappearance of the sensory blockade.
Duration of motor blockade | up to 24 hours
  The duration of motor blockade will be evaluated as the time between the onset of the motor block and the achievement of Grade 0 on the modified Bromage scale.
Motor blockade onset time | During procedure
  The motor blockade onset time will be assessed by movement at the elbow, wrist and fingers using a modified Bromage scale.
Time to need for postoperative first rescue analgesia | During the postoperative 24-hour period.
  The Visual Analogue Scale (VAS) > 3
Consumption of rescue analgesia | During the postoperative 24-hour period.
  The Visual Analogue Scale (VAS) > 3
Postoperative pain | within the first 24 hours (2, 4, 8, 12, 16, and 24 hours).
  Postoperative pain was evaluated with a visual analogue scale